CLINICAL TRIAL: NCT03070704
Title: A Multi-centre, Prospective, Open-label, Single-arm, Non-interventional, Post Marketing Surveillance Study of Xultophy™ (Insulin Degludec/Liraglutide) to Evaluate Long Term Safety and Efficacy in Patients With Type 2 Diabetes Mellitus in Routine Clinical Practice in India
Brief Title: Non-interventional, Post Marketing Surveillance Study of Xultophy™ (Insulin Degludec/Liraglutide) to Evaluate Long Term Safety and Efficacy in Patients With Type 2 Diabetes Mellitus in Routine Clinical Practice in India
Status: Withdrawn | Type: Observational
Why Stopped: Request for the study waived by Indian Health Authorities
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9068-4331; U1111-1185-0871 (Other: WHO)
Record Dates: First submitted 2017-02-24; First posted 2017-03-03 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Insulin degludec /liraglutide
  Interventions: Drug: insulin degludec/liraglutide

INTERVENTIONS:
Drug: insulin degludec/liraglutide — Patients will be treated with commercially available Xultophy™ (insulin degludec / liraglutide) according to routine clinical practice at the discretion of the treating physician

SUMMARY:
This study is conducted in Asia. The aim of this study is to evaluate long term safety and efficacy in patients with type 2 diabetes mellitus in routine clinical practice in India.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are related to the recording of data and determining the suitability for the study according to the protocol. Some specific historical data collected before informed consent is obtained can be used as baseline data (HbA1c, FPG/FBG and others)
* The decision to initiate treatment with commercially available Xultophy™ has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study
* Male or female, age at least 18 years at the time of signing the informed consent
* Patients diagnosed with type 2 diabetes mellitus
* Patients who are scheduled to start treatment with Xultophy™ based on the clinical judgement of their treating physician

Exclusion Criteria:

* Known or suspected hypersensitivity to Xultophy™, any of the active substances, any of the excipients or any related products
* Previous participation in this study. Participation is defined as signed informed consent
* Mental incapacity, unwillingness or language barriers hindering adequate understanding or cooperation
* Females who are pregnant, breast-feeding or intend to become pregnant within the following 12 months
* Patients who are participating in other studies or clinical trials.
* Any disorder which in the opinion of the Physician might jeopardise subject's safety or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on the clinical judgement of their treating physician, patients with type 2 diabetes mellitus will be initiated on Xultophy™ according to routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-08-16 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-08-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent Adverse Events (AEs) | Year 0-1
  Count and % of events

SECONDARY OUTCOMES:
Number of Serious Adverse Events (SAEs) | Year 0-1
  Count and % of events
Number of Serious Adverse Drug Reactions (SADRs) | Year 0-1
  Count and % of events
Number of Adverse Drug Reactions (ADRs) | Year 0-1
  Count and % of events
Number of confirmed hypoglycaemic episodes | Year 0-1
  Count of episodes
Change from baseline in the level of glycosylated haemoglobin (HbA1c) | Year 0, Year 1
  Measured in %
Change in the level of Fasting Plasma/Blood Glucose (FPG/FBG) from baseline | Year 0, Year 1
  Measured in mg/dl or other equivalent SI units
Percentage of patients achieving the target level of HbA1c below 7% | Year 1
  Measured in %
Change in body weight | Year 0, Year 1
  Measured in kg and/or %
Number of patients withdrawn due to ineffective therapy | Year 1
  Count of withdrawals

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com